CLINICAL TRIAL: NCT04395924
Title: Maternal-Foetal Transmission of COVID-19
Brief Title: Maternal-foetal Transmission of SARS-Cov-2
Acronym: TMF-COVID-19
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Collaborators: Centre de Biophysique Moléculaire - Pr Chantal Pichon (Unknown); Professeur TOUMI Hechmi (Unknown)
Responsible Party: Sponsor
Other Study IDs: CHRO-2020-10
Record Dates: First submitted 2020-05-19; First posted 2020-05-20 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-06

CONDITIONS: Maternal Fetal Infection Transmission; COVID-19; SARS-CoV 2
Keywords: Pregnancy; RT-PCR-COVID-19; SARS-CoV 2 serologies; Placenta; Blood cord; Amniotic fluid
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Amniotic fluid, blood cord and placenta.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women COVID-19 positive by RT-PCR: Pregnant women COVID-19 positive by RT-PCR on nasopharyngeal swabs and/or by serology or with previous history of SARS-Cov-2 positive during the pregnancy coming to the maternity to deliver
  Interventions: Diagnostic Test: Diagnosis of SARS-Cov2 by RT-PCR and : IgG, Ig M serologies in the amniotoc fluid, the blood cord and the placenta

INTERVENTIONS:
Diagnostic Test: Diagnosis of SARS-Cov2 by RT-PCR and : IgG, Ig M serologies in the amniotoc fluid, the blood cord and the placenta — During labor and delivery
  1. Sample of amniotic fluid
  2. 2 samples of blood cord after the birth of the new born
  3. 2 samples of placenta
  These samples will be tested with A RT-PCR COVID-19 test and / or serology's A sample of blood cord and placenta will be frozen at -80 degree C and studied for PCR and viral proteome, cytokines , D-dimers and others inflammatory markers in the PRIMMO Laboratory (Prof. TOUMI and LESPESSAILLES) and after in the Centre of molecular biophysics of CNRS of Orleans (Prof. PICHON)

SUMMARY:
One case of maternal-fetal transmission of SARS Cov-2 was published (1). Ig M and Ig G were found at two hours after birth of a new born from a mother COVID-19. Another study on few newborns COVID-19 reported that the SARS-Cov-2 was not transmitted in utero but only after birth.

Although there are few data on COVID-19 during pregnancy, according to our national data collections, it appears to be responsible for miscarriages and fetal deaths. There are also intrauterine growth restrictions and an increase of the rate of cesarean sections for maternal indications. Therefore, it is essential to know if there is a maternal viremia which infects the fetus because the consequences in terms of management would be completely different.

In fact, the potential intrauterine infection will lead to antenatal monitoring of these patients with an antenatal diagnosis and may be a treatment.

Therefore, it seems essential to explore the mode of transmission to the newborn since many newborns have COVID-19 infection The investigators will propose to all pregnant women SARS- Cov-2 positive to perform PCR SARS-Cov-2 tests and /or serology's (IgM and Ig G) on the amniotic fluid, the blood cord and the placenta.

DETAILED DESCRIPTION:
Pregnant women SARS cov-2 positives during pregnancy or during labor tested by a RT-PCR SARS-Cov-2 on nasopharyngeal swabs and/or by serologies.

After informed consent the ivestigators will proceed during labor to:

1. A vaginal swab of amniotic fluid during the rupture of the water pocket during labor.
2. a blood sample from the umbilical cord after delivery of the newborn and clamping and sectioning of the cord. PCR Covid-19 and serologies (Ig M and Ig G) as well as investigating viral proteome and cytokines.

   These are additional samples in addition to the routine samples which have no impact and without risk for the mother the newborn since they are taken after delivery from the side of the placenta after clamping and sectioning of the cord.
3. Samples of 2 fragments of placenta after delivery of the placenta for COVID-19 research, which usually goes to waste or to pathology depending on the clinical context or for infectious tests. In all cases, samples of 3 to 4 cm3 will be taken which will in no way interfere with current analyzes carried out on the placenta which weighs one third of the fetal weight on average. A viral search by COVID-19 PCR will be carried out on the placenta fragment and another part will be frozen for analysis by electron microscopy and study of the viral proteome, cytokines and immune mechanisms. Placenta samples will be frozen at -80 degrees.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women SARS-Cov-2 positive during the pregnancy
* Informed consent obtained
* 18 years to 48 years

Exclusion Criteria:

* Pregnant women without SARS-Cov-2 infection ( PCR test and or serologies negatives)
* curatorship patients.
* Refusal to participate to the study

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women COVID-19 positive or with suspected infection or presented a positive SARS Cov-2 PCR or serologies at any moment of the pregnancy. Symptomatic and asymptomatic pregnant women with SARS-Cov-2 will be included.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-05-05 (Actual); Primary Completion 2021-05-04 (Actual); Study Completion 2021-05-04 (Actual)

PRIMARY OUTCOMES:
COVID-19 by positive PCR in cord blood and / or positive serologies | Day 0
  COVID-19 by positive PCR in cord blood and / or positive serologies

SECONDARY OUTCOMES:
COVID-19 by positive PCR in amniotic fluid and placenta | Day 0
  COVID-19 by positive PCR in amniotic fluid and placenta
New born infected by COVID-19 | Day 0
  Newborn baby infected with COVID-19 on gastric tubing, rectal sample, nasopharyngeal samples by COVID-19 PCR and blood samples by serology

CONTACTS AND LOCATIONS:
Overall Officials: Souhail ALOUINI, M.D., Ph.D., Principal Investigator — CHR ORLEANS
Locations (1):
- CHR Orléans, Orléans, France

REFERENCES:
- [Background] Dong L, Tian J, He S, Zhu C, Wang J, Liu C, Yang J. Possible Vertical Transmission of SARS-CoV-2 From an Infected Mother to Her Newborn. JAMA. 2020 May 12;323(18):1846-1848. doi: 10.1001/jama.2020.4621. PMID 32215581
- [Background] Sutton D, Fuchs K, D'Alton M, Goffman D. Universal Screening for SARS-CoV-2 in Women Admitted for Delivery. N Engl J Med. 2020 May 28;382(22):2163-2164. doi: 10.1056/NEJMc2009316. Epub 2020 Apr 13. No abstract available. PMID 32283004
- [Background] Wang W, Xu Y, Gao R, Lu R, Han K, Wu G, Tan W. Detection of SARS-CoV-2 in Different Types of Clinical Specimens. JAMA. 2020 May 12;323(18):1843-1844. doi: 10.1001/jama.2020.3786. PMID 32159775
- [Background] Woo PC, Lau SK, Wong BH, Tsoi HW, Fung AM, Chan KH, Tam VK, Peiris JS, Yuen KY. Detection of specific antibodies to severe acute respiratory syndrome (SARS) coronavirus nucleocapsid protein for serodiagnosis of SARS coronavirus pneumonia. J Clin Microbiol. 2004 May;42(5):2306-9. doi: 10.1128/JCM.42.5.2306-2309.2004. PMID 15131220